CLINICAL TRIAL: NCT00953654
Title: Exercise Training for the Treatment of Generalized Anxiety Disorder: A Randomized Controlled Trial Comparing Endurance and Strength Training Among Sedentary Women With Generalized Anxiety Disorder.
Brief Title: Exercise Training for the Treatment of Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UGA-2009-01913-1
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2010-09-29 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-07

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Exercise Training; Strength Training; Mental Health
MeSH Terms: conditions — Generalized Anxiety Disorder; Psychological Well-Being | interventions — Resistance Training; Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Strength Training (Experimental): Lower-body strength training exercise twice weekly for 6 weeks at an intensity progressing from 50% to 75% predicted one-repetition maximum
  Interventions: Other: Strength Training
- Endurance Training (Experimental): Six-week lower-body dynamic cycling exercise condition completed twice weekly and matched to the strength training arm on total work completed, total time actively engaged in exercise and load progression.
  Interventions: Other: Endurance Training
- Waiting List Control (No Intervention): Waiting list control condition in which participants will maintain their current lifestyle and will not enter a six-week exercise training intervention, but will complete outcome measures along the same time progression as the intervention arms.

INTERVENTIONS:
Other: Strength Training — 6 weeks of strength training exercise sessions involving leg press, leg curl, and leg extension exercises twice weekly at an intensity progressing from 50% to 75% of predicted one-repetition maximum across the 6 weeks of the trial.
  Arms: Strength Training
Other: Endurance Training — Six weeks of lower-body dynamic cycling exercise completed on an electronically-braked cycle ergometer twice weekly. The intervention will be matched to the strength training intervention on total work completed, total time actively engaged in exercise, a focus on leg muscles, and load (intensity) progression across the 6 week training protocol.
  Arms: Endurance Training

SUMMARY:
The purpose of this study is to compare the effects of 6 weeks of endurance or strength training and a wait list comparison condition on symptoms of Generalized Anxiety Disorder (GAD).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-39 years
* Principal diagnosis of Generalized Anxiety Disorder according to DSM-IV diagnostic criteria (comorbidities will be acceptable as long as Generalized Anxiety Disorder is the principal diagnosis)

Exclusion Criteria:

* A score of less than 45 on the Penn State Worry Questionnaire
* A score of less than 7 on the Generalized Anxiety Disorder section of the Psychiatric Diagnostic Screening Questionnaire
* Expending greater than 250 kilocalories per kilogram body weight per week as measured by a 7-day physical activity recall questionnaire
* Engaging in greater than 6 exercise bouts in the month prior to recruitment
* Pregnancy
* Any medical contraindications (cardiovascular or musculoskeletal) to exercise training according to American College of Sports Medicine guidelines

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew P Herring, MS, MEd, Principal Investigator — The University of Georgia; Patrick J O'Connor, PhD, Study Director — The University of Georgia
Locations (1):
- The University of Georgia, Athens, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were recruited from from a University and Community setting from August 2009 to March 2010. 1044 women were screened using online screening questionnaires; 853 were excluded for having too few worry symptoms or too high a physical activity level. 55 completed diagnostic interviews - 25 were excluded for no Generalized Anxiety Disorder.
Pre-assignment Details: Thirty women met exclusion criteria and were enrolled in the trial.
Groups:
- Resistance Exercise Training: Lower-body strength training exercise twice weekly for 6 weeks at an intensity progressing from 50% to 75% predicted one-repetition maximum
- Aerobic Exercise Training: Six-week dynamic leg cycling exercise condition completed twice weekly and matched to the strength training arm on total positive work completed, total time actively engaged in exercise and weekly load progression.
Period: Overall Study
Arm/Group | Resistance Exercise Training | Aerobic Exercise Training | Waiting List Control
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistance Exercise Training | Aerobic Exercise Training | Waiting List Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Customized [Number; unit: participants]
  ≥18 and ≤23 years | 6 | 8 | 6 | 20
  >23 and ≤29 years | 1 | 2 | 1 | 4
  >29 and ≤37 years | 3 | 0 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (7.1) | 20.7 (3.0) | 24.2 (6.3) | 23.5 (5.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 10 | 10 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 30
Psychiatric Comorbidity [Number; unit: cases] — Number of comorbid psychiatric diagnoses was assessed using the Adult Version of the Anxiety Disorders Interview Schedule for the DSM-IV (ADIS-IV).
  cases
    Specific Phobia | 2 | 5 | 10 | 17
    Social Phobia | 2 | 5 | 5 | 12
    Obsessive Compulsive Disorder (OCD) | 1 | 1 | 3 | 5
    Post-Traumatic Stress Disorder (PTSD) | 0 | 0 | 2 | 2
    Major Depressive Disorder (MDD) | 1 | 3 | 3 | 7
    Dysthymia | 2 | 0 | 2 | 4
    Substance Abuse | 1 | 0 | 0 | 1
Medication [Number; unit: Participants] — Non-psychoactive and psychoactive medication use was assessed by self-report using a medication use recall questionnaire.
  Participants
    Contraceptive | 5 | 5 | 5 | 15
    Selective Serotonin Reuptake Inhibitor (SSRI) | 2 | 2 | 3 | 7
    Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) | 1 | 1 | 0 | 2
    Norepinephrine-Dopamine Reuptake Inhibitor (NDRI) | 0 | 1 | 1 | 2
    Muscle Relaxant | 1 | 1 | 0 | 2
    Psychostimulant | 0 | 0 | 1 | 1
    Antibiotic | 0 | 1 | 0 | 1
    Antihistamine | 1 | 0 | 0 | 1
Weight [Mean (Standard Deviation); unit: Kilograms] | 60.6 (9.1) | 70.0 (15.5) | 66.4 (8.1) | 65.7 (12.2)
Height [Mean (Standard Deviation); unit: centimeters] | 162.6 (6.2) | 165.0 (7.6) | 166.5 (4.6) | 164.7 (6.6)

OUTCOME MEASURES:

1. Primary Outcome: Generalized Anxiety Disorder (GAD) Remission as Measured by Anxiety Disorders Interview Schedule-Adult Version (ADIS-IV) Severity Ratings
Description: GAD is characterized by persistent excessive or pathologic worry most days for at least 6 months about activities of daily life that is difficult to control and associated with at least 3 of the following symptoms: restlessness, feeling on edge, being easily fatigued, difficulty concentrating, irritability, muscle tension, and sleep difficulty. Symptoms are not caused by a substance or disorder, but cause significant distress or functional impairment. Remission was measured using the ADIS-IV from 1-16 days following the 6-week intervention.
Time Frame: Pre- and post- 6 week training intervention
Measure: Number; unit: Participants
Arm/Group | Resistance Exercise Training | Aerobic Exercise Training | Waiting List Control
Number analyzed (Participants) | 10 | 10 | 10
Participants | 4 | 6 | 7

2. Primary Outcome: Worry Symptoms
Description: Worry symptoms, hallmark symptoms of GAD, were assessed using the Penn State Worry Questionnaire (PSWQ). The PSWQ is a 16-item self-report questionnaire that measures pathological worry symptoms. Participants rate items from 1 "not at all typical of me" to 5 "very typical of me." Scores range from 16 to 80, with higher scores indicated exacerbated worry symptoms. Symptoms were assessed at baseline and at the beginning of the second weekly session during weeks 2, 4, and 6.
Time Frame: Baseline, Week 2, Week 4, Week 6
Measure: Mean (Standard Deviation); unit: Units on a scale (PSWQ)
Units Other Than Participants: Units on a scale
Arm/Group | Resistance Exercise Training | Aerobic Exercise Training | Waiting List Control
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (Units on a scale) | 16 | 16 | 16
Units on a scale (PSWQ)
  Baseline | 63.80 (9.78) | 62.1 (6.4) | 64.3 (7.01)
  Week 2 | 59.83 (9.93) | 63.20 (4.16) | 63.4 (8.91)
  Week 4 | 60.3 (8.29) | 58.8 (5.2) | 63.5 (7.04)
  Week 6 | 61.1 (10.01) | 59.3 (7.38) | 65.5 (7.62)
Statistical Analysis 1: Comparison: Resistance Exercise Training vs Aerobic Exercise Training vs Waiting List Control; Effects of RET and AET were compared to WL using a 3 condition by 3 time ANCOVA. An a priori statistical power analysis showed that a sample of 30 patients would provide a statistical power of .80 to detect a condition-by-time interaction for PSWQ scores assuming a two-tailed alpha value of 0.05, a correlation across repeated measures of 0.75 and a desire to detect a standardized effect size of 0.65; Test type: Superiority or Other; p < 0.05, ANCOVA; The degrees of freedom were adjusted when the sphericity assumption was violated based on Mauchly's test

ADVERSE EVENTS:
Time Frame: Across 6-week intervention
Description: Adverse events including any musculoskeletal injuries or increases in suicidal ideation (measured with ninth item of Beck Depression Inventory-II) were monitored for each patient during each week of the 6-week intervention.
Arm/Group | Resistance Exercise Training | Aerobic Exercise Training | Waiting List Control
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
One limitation of this trial was the small sample size. Although the research design was sufficiently powered to detect a statistically significant effect for the primary outcome, a larger trial is warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes